CLINICAL TRIAL: NCT03405636
Title: Prospective, Non-randomized, Open Label Clinical Study to Assess the Safety and Performance of the Xeltis Pulmonary Valved Conduit in Subjects Undergoing Right Ventricular Outflow Tract (RVOT) Reconstruction
Brief Title: Xeltis Pulmonary Valved Conduit Safety and Performance Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not started
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-02
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xeltis Pulmonary Valved Conduit (Experimental): PV Conduit for RVOT reconstruction
  Interventions: Device: Xeltis Pulmonary Valved Conduit

INTERVENTIONS:
Device: Xeltis Pulmonary Valved Conduit — RVOT reconstruction

SUMMARY:
This is a multi-center prospective, single-arm, non-randomized, open label study to assess safety and performance of the Xeltis Pulmonary Valved Conduit in subjects requiring Right Ventricular Outflow Tract correction or reconstruction due to congenital heart malformations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring RVOT reconstruction, suitable for 16 mm or 18 mm valved conduit.
2. Male or Female.
3. Age < 22 years.
4. Right Ventricular to Pulmonary Artery mean gradient > 35mm Hg or moderate or severe Pulmonary regurgitation (≥3+), or have both.
5. The patient, and the patient's parent / legal representative where appropriate, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent by signing the approved informed consent form.
6. The patient, and the patient's parent / legal representative where appropriate, and the treating physician agree that the subject will return for all required post-procedure follow up visits and the subject will comply with clinical investigation plan required follow-up visits.

Exclusion Criteria:

1. Need for or presence of prosthetic heart valve at other position
2. Need for concomitant surgical procedures (non-cardiac)
3. Patients with previously implanted pacemaker (including defibrillators) or mechanical valves
4. Active bacterial or viral infection or requiring current antibiotic therapy (if temporary illness, patient may be a candidate 4 weeks after discontinuation of antibiotics)
5. Active endocarditis
6. Leukopenia, according to local laboratory evaluation of white blood cell count
7. Acute or chronic anemia, according to local laboratory evaluation of hemoglobin Patients can be transfused to meet eligibility criteria
8. Thrombocytopenia, defined as Platelet count < 150,000/mm3 Patients can be transfused to meet eligibility criteria
9. Severe chest wall deformity, which would preclude placement of the PV conduit
10. Pulmonary hypertension (right ventricular systolic pressure ≥ half of systemic systolic pressure)
11. Right ventricular outflow tract aneurysm
12. Known hypersensitivity to anticoagulants and antiplatelet drugs and to the device materials
13. Immunocompromised patient defined as: autoimmune disease, patients receiving immunosuppressant drugs or immune stimulant drugs
14. Patient has chronic inflammatory / autoimmune disease
15. Need for emergency cardiac or vascular surgery or intervention
16. Major or progressive non-cardiac disease (liver failure, renal failure, cancer) that has a life expectancy of less than one year
17. Currently participating, or participated within the last 30 days, in an investigational drug or device study
18. Alcohol or drug abuse as defined by DSM IV-TR criteria for substance abuse - this includes the illicit use of cannabis within the last 12 months
19. Females who are sexually active and are not willing to use adequate contraceptive precautions for the next 2 years
20. Patient has medical, social or psychosocial factors that, in the opinion of the Investigator, could have impact on safety or compliance

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Survival at 12 months follow up post implantation | 12 months
  Measured by the fact that the patient is still alive at the time of the 12 month FU visit

SECONDARY OUTCOMES:
Freedom from device related death, intervention and/or reoperation at 12 months follow up | 12 months
  Measured by the fact that the patient did not die, did not have a reoperation or reintervention during the first 12 months
Mean pressure gradient across the area of conduit implantation (RV to PA) of less than 40 mm Hg at 12 months follow up | 12 months
Pulmonary regurgitation of equal or less than moderate (≤40 %) at 12 months follow up | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Gottsegen György Hungarian Institute of Cardiology, Paediatric Cardiac Centre, Budapest, Hungary
- Institute Jantung Negara, National Heart Institute, Kuala Lumpur, Malaysia
- University Children's Hospital of Cracow (UCH),, Krakow, Poland
- Childrens Heart Centre Slovak Republic, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No